CLINICAL TRIAL: NCT01470157
Title: A Randomized, Clinical Trial of Oral Midazolam Plus Placebo Versus Oral Midazolam Plus Oral Ketamine for Sedation During Laceration Repair
Brief Title: A Clinical Trial of Oral Midazolam Plus Oral Ketamine for Sedation During Laceration Repair
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Director, Pediatric Emergency Unit, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22/11
Record Dates: First submitted 2011-09-19; First posted 2011-11-11 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Lacertaions
MeSH Terms: interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): Oral Ketamine in addition to oral midazolam
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Normal saline (placebo) in addition to oral midazolam
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Ketamine — 5mg/kg as oral suspension
  Arms: Ketamine
Drug: Normal Saline — Normal Saline (placebo) in addition to Midazolam 0.5mg/kg as oral suspension
  Arms: Placebo

SUMMARY:
Background: Sedation is often needed for young children undergoing minor procedures in the emergency department (ED). Oral midazolam is one of the most commonly used regimens for children undergoing laceration repair but its sedative efficacy was shown to be suboptimal. In a few studies oral ketamine has been used successfully for procedural sedation as well. The efficacy of using a combination of oral midazolam and oral ketamine for procedural sedation has been studied only for invasive procedures in children with malignancies. No randomized controedll studies were performed using this sedative combination in children requiring laceration repair. Objectives: To determine the efficacy of adding oral ketamine to oral midazolam for procedural sedation in children requiring laceration repair compares to oral midazolam plus placebo. Design: A randomized, double blind, placebo-controlled study. Setting: Pediatric Emergency Department. Participants: Children 1 to 10 years with laceration requiring sedation. Interventions: Eligible patients will be randomly assigned to one of two treatment groups: oral midazolam plus oral placebo group and oral midazolam plus oral ketamine group. Both groups will be given the same volume of medications. Midazolam will be given orally in a dose of 0.5 mg/kg (max.-15 mg) with placebo or 0.5 mg/kg (max.- 15 mg) with oral ketamine in a dose of 5 mg/kg. The medical staff will be blinded to the treatment given. Patient monitoring will be conducted according to the American Academy of Pediatrics (APP) and the Israeli health ministry guidelines for monitoring and management of pediatric patients during and after sedation for diagnostic and therapeutic procedures. Main outcome measures: Pain score: Visual Analog Score (VAS) - by parent. Data analysis: Descriptive statistics will be used to describe the study population. Data will be analyzed using t- tests for continuous data and Fisher exact test for categorical data.

Key words: sedation, children, ketamine, midazolam, emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Age: 1 years - 10 years
* Any child with laceration requiring sedation

Exclusion Criteria:

* Major trauma
* Closed head injury associated with loss of consciousness
* Abnormal neurologic examination in a previously normal child
* Significant developmental delay or baseline neurological deficit
* A patient with seizures
* Elevated intra-cranial pressure
* Hypersensitivity to midazolam or ketamine
* Hypertension
* Hyperthyroidism or a patient receiving thyroid replacement
* alcohol intoxication or a history of alcohol abuse
* Acute or chronic respiratory, cardiac, renal or hepatic abnormalities
* Glaucoma
* Known psychiatric disease
* ASA score of more than 2
* Informed consent cannot be obtained from legal guardian

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-03 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Pain score: Visual analog score (VAS)- by parent | participants will be followed for the duration of hospital stay, an expected average of 3 hours

SECONDARY OUTCOMES:
Pain score: Visual analog score (VAS)- by a physician | while in the ED for about 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Emergency Department, Assaf Harofeh, Zerifin, Israel

REFERENCES:
- [Derived] Barkan S, Breitbart R, Brenner-Zada G, Feldon M, Assa A, Toledano M, Berkovitch S, Shavit I, Kozer E. A double-blind, randomised, placebo-controlled trial of oral midazolam plus oral ketamine for sedation of children during laceration repair. Emerg Med J. 2014 Aug;31(8):649-53. doi: 10.1136/emermed-2012-202189. Epub 2013 May 18. PMID 23686730